CLINICAL TRIAL: NCT07163819
Title: Effect of Probiotic Intervention on Travel-Related Health Conditions During Short-Term Overseas Travel
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Tsinghua University Science and Technology (Unknown)
Responsible Party: Principal Investigator, Min-Tze LIONG, Prof., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: THU-01-2025-1007
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adults
Keywords: probiotic; international travel
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Daily 6-drops of non-GMO corn starch in medium-chain triglyceride oil
  Interventions: Other: Placebo
- Probiotic (Experimental): Daily 6-drops of Bifidobacterium longum subsp. infantis M-63, B. breve M-16V, and B. longum BB536 in non-GMO corn starch as excipient, in medium-chain triglyceride oil (1.5 × 109 CFU/day)
  Interventions: Other: Probiotic

INTERVENTIONS:
Other: Probiotic — Daily 6-drops of Bifidobacterium longum subsp. infantis M-63, B. breve M-16V, and B. longum BB536 in non-GMO corn starch as excipient, in medium-chain triglyceride oil (1.5 × 109 CFU/day)
  Arms: Probiotic
Other: Placebo — Daily 6-drops of non-GMO corn starch in medium-chain triglyceride oil
  Arms: Placebo

SUMMARY:
International travel disrupts gut health through dietary changes, microbial exposure, and stress, often causing gastrointestinal symptoms like traveler's diarrhea and sleep disturbances. These shifts may increase antibiotic resistance risks. Probiotics may help stabilize gut microbiota and improve well-being during travel. This randomized, double-blind, placebo-controlled trial investigated whether probiotic supplementation mitigates gut microbiota perturbations, gastrointestinal symptoms, and sleep issues in adults traveling abroad. The investigators also assessed changes in anxiety, well-being, gut immunity, microbial function, and antibiotic resistance genes.

DETAILED DESCRIPTION:
International travel exposes individuals to abrupt changes in diet, water sources, microbial exposures, sleep schedules, and psychological stress. These factors often perturb the gut microbiota and influence host health outcomes. Studies have reported significant fluctuations in gut microbiota among travelers, even in those without diarrheal symptoms, with marked shifts in microbiome composition during short-term travel. Such perturbations are frequently accompanied by gastrointestinal symptoms and reduced well-being, highlighting the need for strategies to maintain gut homeostasis during travel.

Traveler's diarrhea remains one of the most common travel-related illnesses, with incidence rates varying from 30-70% depending on destination and season. Gastrointestinal discomfort during travel extends beyond diarrhea to include abdominal pain, abnormal gut transit, loose stools, and other non-diarrheal symptoms. These issues can significantly impact travel comfort and enjoyment.

International travel has also been associated with increased risk of acquiring antimicrobial-resistant organisms and genes, posing concerns for both individual and public health. The gut environment facilitates the selection and exchange of antibiotic resistance determinants, with studies showing increased abundance and diversity of antimicrobial resistance genes following travel.

Sleep disturbances represent another significant challenge during travel, arising from time zone changes and adaptation to new environments. These disruptions can profoundly affect well-being given sleep's critical role in health. The relationship between sleep and gut microbiota through the microbiome-gut-brain axis suggests that sleep disturbances during travel may contribute to gastrointestinal vulnerability through neuroendocrine, immune, and metabolic pathways.

Probiotics, defined as live microorganisms that confer health benefits when administered in adequate amounts, represent a potential intervention strategy. Evidence suggests probiotics enhance colonization resistance against pathogens, modulate immune responses, strengthen epithelial barrier integrity, and generate beneficial metabolites. Beyond gastrointestinal benefits, probiotics may influence systemic inflammation, lipid metabolism, and mental health outcomes through the gut-brain axis. While some evidence supports their role in reducing gastrointestinal transit time and constipation symptoms, as well as modest protection against traveler's diarrhea, robust data specifically regarding travel-related probiotic interventions remains limited.

The investigators conducted a randomized, double-blind, placebo-controlled trial in healthy adults undertaking short-term international travel. The study aimed to determine whether daily probiotic supplementation attenuates travel-associated perturbations in gut microbiota composition and diversity, while assessing concurrent changes in gastrointestinal symptoms, sleep quality, anxiety, and subjective well-being using validated instruments. Functional outcomes included assessment of specific microbial species, secretory immunoglobulin A, vitamin-related indices, antibiotic resistance genes, and metabolic pathway analyses to provide mechanistic insights. The investigators hypothesized that probiotic supplementation would stabilize the gut microbiota, enrich beneficial taxa and functions, and improve both gastrointestinal comfort and psychological outcomes compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy adults
* Scheduled to undertake a short-term round trip (less than 7 days) to abroad
* Able to complete study procedures
* Willing to take intervention products

Exclusion Criteria:

* Use of antibiotics, probiotics, hormones, immunosuppressants, biologics or JAK inhibitors within four weeks prior to study
* Chronic or severe systemic diseases (including cardiovascular, hepatic, renal, malignant or psychiatric disorders)
* Uncontrolled parasitic infections
* Long-term use of corticosteroids, growth hormone, vitamin B12, lysine or inositol
* Major surgery within one month
* Allergy to probiotic components
* Other conditions deemed inappropriate by investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiota profiles of fecal samples in generally healthy adults upon administration of probiotic as assessed via metagenomics sequencing | 7 days
  Differences in microbiota abundance in fecal sample of generally healthy adults upon administration o probiotic compared to placebo

SECONDARY OUTCOMES:
Respiratory symptoms duration and frequency in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Changes in duration and frequency of respiratory illnesses symptoms from generally healthy adults on probiotic or placebo after 7-days, via the use of standard clinical assessment questionnaire, scale 0-3 where higher scores indicate more severe symptoms.
Gastrointestinal symptoms in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in duration and frequency of gastrointestinal symptoms upon administration of probiotic compared to placebo via the use of standard clinical assessment questionnaire, scale 0-3 where higher scores indicate more severe symptoms.
Allergy symptoms in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in duration and frequency of allergy symptoms upon administration of probiotic compared to placebo via the use of standard clinical assessment questionnaire, scale 0-3 where higher scores indicate more severe symptoms.
Gastrointestinal metabolites in generally healthy adults upon administration of probiotic as assessed using LC-MS | 7 days
  Differences in concentrations of gastrointestinal metabolites upon administration of probiotic compared to placebo
Quality of life in generally healthy adults upon administration of probiotic as assessed using questionnaire | 7 days
  Differences in quality of life via the use of questionnaires such as anxiety (GAD-7, scale 0-3 where higher scores indicate more severe outcomes), sleep (PSQI, scale 0-3 where higher scores indicate more severe outcomes) and well-being (WHO-5, scale 0-5 where higher scores indicate better outcomes) upon administration of probiotic compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Ai Zhou, Ph.D., Principal Investigator — Tsinghua University Science and Technology
Locations (2):
- Tsinghua University Science and Technology, Haidian, Beijing Municipality, China
- Universiti Sains Malaysia, George Town, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No